CLINICAL TRIAL: NCT05912712
Title: Safety And Efficacy Study of Autologous Platelet-rich Plasma (PRP) and Thrombin Coagulum for the Topical Treatment of Rectal Mucosal Ulcers
Brief Title: Autologous Platelet-rich Plasma (PRP) and Thrombin Coagulum for the Topical Treatment of Rectal Mucosal Ulcers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Jie Liang, Professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XijingHDD-UC-PG
Record Dates: First submitted 2023-05-15; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Ulcerative Colitis Chronic Moderate; Ulcerative Colitis Chronic Severe; Rectal Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Platelet-rich Plasma (PRP) Gel Treatment Group (Experimental): Rectal 10ml platelet rich plasma gel enema + infliximab standard treatment at fixed time every day for seven consecutive days
  Interventions: Other: Autologous Platelet-rich Plasma (PRP) and Thrombin Coagulum Treatment; Biological: Infliximab Treatment
- Platelet Poor Plasma (PPP) Gel Treatment Group (Sham Comparator): Rectal 10ml PPP gel enema + infliximab standard treatment for 7 consecutive days
  Interventions: Other: Autologous Platelet-poor Plasma (PPP) and Thrombin Coagulum Treatment; Biological: Infliximab Treatment
- Mesalazine Suppository Treatment Group (Active Comparator): Patients were given 1g mesalazine suppository and infliximab daily for 7 consecutive days
  Interventions: Drug: Mesalazine Suppository Treatment; Biological: Infliximab Treatment

INTERVENTIONS:
Other: Autologous Platelet-rich Plasma (PRP) and Thrombin Coagulum Treatment — 10 mL PRP and thrombin coagulum gel was administered every night for seven consecutive days by the same IBD specialist. Before the intervention, the patients had to defecate. The prepared PRP gel was injected into the external opening of the rectum using the same syringe, and the patient was kept in the Trendelenburg position to ensure that the therapeutic drug remained in place under gravity. The normal supine position was returned after 15 minutes to minimize PRP leakage. The outflow was observed, and the amount of outflow was recorded.
  Arms: Platelet-rich Plasma (PRP) Gel Treatment Group
Other: Autologous Platelet-poor Plasma (PPP) and Thrombin Coagulum Treatment — 10 mL PPP and thrombin coagulum gel was administered every night for seven consecutive days by the same IBD specialist. Before the intervention, the patients had to defecate. The prepared PPP gel was injected into the external opening of the rectum using the same syringe, and the patient was kept in the Trendelenburg position to ensure that the therapeutic drug remained in place under gravity. The normal supine position was returned after 15 minutes to minimize PPP leakage. The outflow was observed, and the amount of outflow was recorded.
  Arms: Platelet Poor Plasma (PPP) Gel Treatment Group
Drug: Mesalazine Suppository Treatment — For patients receiving mesalazine suppositories, the intervention was inserted through the anus with a disposable sanitary finger to the point of slight loss of resistance. To facilitate intervention, moisturize with water or cream. If the drug drains within 10 minutes, it should be re-inserted. The swelling at the local injection site on each group's intervention day was recorded.
  Arms: Mesalazine Suppository Treatment Group
Biological: Infliximab Treatment — Patients, in every arm, all receive infliximab (300 mg iv at 0, 2, 6 weeks, and then every eight weeks).

SUMMARY:
Ulcerative colitis (UC) is a chronic persistent inflammatory disease. The lesions are mainly confined to the large intestine and continuously affect the rectum and part or all of the colon. Its histological characteristics are diffuse neutrophil infiltration in the lamina propria of the colon mucosa, mucosal erosion, ulcer, cryptitis, and crypt abscess. The most common clinical manifestations are abdominal pain, diarrhea, and bloody mucopurulent stool, accompanied by extraintestinal manifestations such as mouth, skin, joints, and eyes. Severe lesions can be complicated by toxic megacolon, intestinal perforation, lower gastrointestinal hemorrhage, intraepithelial neoplasia, and cancer, so surgical treatment is necessary. Studies have reported that UC patients have a 10-year cumulative recurrence risk of 70%-80%, nearly 50% of patients require UC-related hospitalization, and the 5-year risk of re-hospitalization is ~ 50%. The 5-year and 10-year cumulative risk of patients undergoing colectomy is 10%-15%, which dramatically endangers the health of patients and reduces the quality of life of patients.

Currently, the commonly used medical treatment drugs for UC patients include 5-aminosalicylic acid, topical and systemic glucocorticoids, immunomodulators, anti-tumor necrosis factor drugs, and other biological agents. The most commonly used optimization methods are drug escalation therapy and combining drugs with different mechanisms. The real-world data results of an initial population-based cohort study from six Asian countries showed that the endoscopic mucosal healing rate of patients with ulcerative colitis in the first year of diagnosis was 38.2%, and the histological mucosal healing rate was 23.1%. It can be expected that the mucosal healing rate of patients with moderate to severe UC may be lower. Long-term chronic recurrent diseases may lead to poorer quality of life, extended hospital stays, heavier financial burdens, and more physical and mental pain. Therefore, optimizing the treatment plan for patients with moderate to severe UC needs more exploration and research.

Autologous Platelet-rich plasma (A-PRP) is A platelet-rich concentrate obtained by centrifugation of whole blood. As a concentrated source of autologous platelets, they contain a large number of Growth factors (GF) and cytokines, such as platelet-derived Growth factor (PDGF), transforming growth factor β(TGF-β), vascular endothelial growth factor (VEGF) and epithelial growth factor (EGF), which regulate cell function. Such as attachment, macrophage migration, proliferation, and differentiation, promote extracellular matrix accumulation and ultimately improve tissue healing and regeneration. At the same time, A-PRP has A lower risk of adverse reactions such as immune rejection and allergy due to its isolation from autologous blood.

After PRP is induced by activators such as calcium and thrombin, activated platelets degranulate immediately and secrete multiple high concentrations of growth factors. 70% of the growth factors can be released within 10 minutes of activation, and more than 95% can be released within the first hour. Platelet-rich Gel (PG), which can embed growth factors to improve clinical efficacy, keeps platelets and their release products in the target wound area and promotes healing.

Although the safety and efficacy of PRP still need to be fully confirmed by large-scale clinical trials, its sound effect has been verified in many clinical practices and basic scientific research in cell culture and animal models. At present, it mainly includes the treatment of oral and maxillofacial external, musculoskeletal system, plastic skin, and chronic wounds (such as pressure ulcers, venous leg ulcers, diabetic foot ulcers, etc.). They can be mixed into bone grafts, sprayed on soft tissue surfaces as a biofilm, or made into eye drops.

The use of PRP in intestinal mucosal ulcers has rarely been reported. There are no prospective randomized studies of its clinical use in patients with ulcerative colitis. Therefore, we planned to conduct a prospective, randomized, double-blind, controlled clinical trial to investigate the efficacy and safety of repeated treatment with autologous platelet-rich plasma gel on an intestinal mucosal ulcer in patients with moderate to severe UC involving the rectum in Xijing Hospital, China IBD Regional Center. To provide a new option for remission induction therapy in patients with moderate to severe ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

1. Platelet ≥150×10^9g/L, hemoglobin ≥60g/L;
2. Patients with ulcerative colitis were diagnosed according to the diagnostic criteria of ulcerative colitis in the 2018 China's National consensus on the diagnosis and treatment of inflammatory bowel disease;
3. Patients with moderate to severe ulcerative colitis involving the rectum or refractory distal rectal ulcerative colitis (modified Mayo score ≥6 and endoscopic Mayo score ≥2);
4. Patients with ulcerative colitis who were initially treated with infliximab (according to a regular intravenous infusion schedule of 0w, 2w, 6w, and then every 8w);
5. Patients who were able and willing to adhere to the study protocol provided signed, dated, written informed consent.

Exclusion Criteria:

1. Patients with platelet-related bleeding diseases (such as Henoch-Schonlein purpura, coagulopathy, primary/secondary thrombocytopenia, etc.);
2. Medications with anticoagulant effects such as nonsteroidal anti-inflammatory drugs, heparin, coumarin, warfarin, aspirin, etc. (acetaminophen was used to treat discomfort during the study period);
3. Patients using mesalazine enema solution during treatment;
4. Patients with active infection of intestinal or other extra-intestinal organs (hepatitis, active tuberculosis, etc.);
5. Patients with known hypersensitivity to calcium gluconate and thrombin
6. Patients who may require immediate surgical treatment;
7. Pregnant or nursing mothers;
8. Patients with severe liver and kidney dysfunction, heart failure or other serious systemic diseases;
9. Any conditions that prevent the completion of the study or interfere with the analysis of the study results, including drug or alcohol abuse history, smoking abstinence, mental illness or poor compliance, and clear immune system (including HIV infection), blood system or cancer related diseases;
10. Patients who withdraw consent;
11. Patients enrolled in other clinical trials within 3 months prior to screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Endoscopic response rate of local treatment with autologous platelet-rich plasma gel | 14 weeks
  Endoscopic response rate of local treatment with autologous platelet-rich plasma gel in patients with moderate to severe ulcerative colitis involving the rectum.

SECONDARY OUTCOMES:
Endoscopic remission rate of local treatment with autologous platelet-rich plasma gel | 1 week and 14 weeks
  Endoscopic remission rate of local treatment with autologous platelet-rich plasma gel in patients with moderate to severe ulcerative colitis involving the rectum.
Clinical response rate of PRP-thrombin coagulum treatment on Rectal Mucosal Ulcers | 1 week and 14 weeks
  The clinical response rate will be analyzed.
Clinical remission rate of PRP-thrombin coagulum treatment on Rectal Mucosal Ulcers | 1 week and 14 weeks
  The clinical remission rate will be analyzed.
Inflammatory parameter alteration with PRP-thrombin coagulum treatment on Rectal Mucosal Ulcers | 1 week, 2 weeks, 6 weeks, and 14 weeks
  The erythrocyte sedimentation rate will be analyzed.
Inflammatory response alteration with PRP-thrombin coagulum treatment on Rectal Mucosal Ulcers | 1 week, 2 weeks, 6 weeks, and 14 weeks
  The C-reactive protein concentration will be analyzed.
Incidence of Adverse Events | 1 week, 2 weeks, 6 weeks, and 14 weeks
  Adverse events will reported at the start and throughout the treatment period.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Digestive Disease, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fumery M, Singh S, Dulai PS, Gower-Rousseau C, Peyrin-Biroulet L, Sandborn WJ. Natural History of Adult Ulcerative Colitis in Population-based Cohorts: A Systematic Review. Clin Gastroenterol Hepatol. 2018 Mar;16(3):343-356.e3. doi: 10.1016/j.cgh.2017.06.016. Epub 2017 Jun 16. PMID 28625817
- [Background] Leung CM, Tang W, Kyaw M, Niamul G, Aniwan S, Limsrivilai J, Wang YF, Ouyang Q, Simadibrata M, Abdullah M, Ong DE, Yu HH, Zhang J, Ching J, Wu JCY, Chan FKL, Sung JJY, Ng SC. Endoscopic and Histological Mucosal Healing in Ulcerative Colitis in the First Year of Diagnosis: Results from a Population-based Inception Cohort from Six Countries in Asia. J Crohns Colitis. 2017 Dec 4;11(12):1440-1448. doi: 10.1093/ecco-jcc/jjx103. PMID 28961760
- [Background] Lee JW, Kwon OH, Kim TK, Cho YK, Choi KY, Chung HY, Cho BC, Yang JD, Shin JH. Platelet-rich plasma: quantitative assessment of growth factor levels and comparative analysis of activated and inactivated groups. Arch Plast Surg. 2013 Sep;40(5):530-5. doi: 10.5999/aps.2013.40.5.530. Epub 2013 Sep 13. PMID 24086805
- [Background] Lee JH, Kim MJ, Ha SW, Kim HK. Autologous Platelet-rich Plasma Eye Drops in the Treatment of Recurrent Corneal Erosions. Korean J Ophthalmol. 2016 Apr;30(2):101-7. doi: 10.3341/kjo.2016.30.2.101. Epub 2016 Mar 25. PMID 27051257
- [Background] Marx RE. Platelet-rich plasma: evidence to support its use. J Oral Maxillofac Surg. 2004 Apr;62(4):489-96. doi: 10.1016/j.joms.2003.12.003. No abstract available. PMID 15085519
- [Background] Nikolidakis D, Jansen JA. The biology of platelet-rich plasma and its application in oral surgery: literature review. Tissue Eng Part B Rev. 2008 Sep;14(3):249-58. doi: 10.1089/ten.teb.2008.0062. PMID 18601587
- [Background] Al-Hamed FS, Abu-Nada L, Rodan R, Sarrigiannidis S, Ramirez-Garcialuna JL, Moussa H, Elkashty O, Gao Q, Basiri T, Baca L, Torres J, Rancan L, Tran SD, Lordkipanidze M, Kaartinen M, Badran Z, Tamimi F. Differences in platelet-rich plasma composition influence bone healing. J Clin Periodontol. 2021 Dec;48(12):1613-1623. doi: 10.1111/jcpe.13546. Epub 2021 Sep 27. PMID 34517437
- [Background] Hesseler MJ, Shyam N. Platelet-rich plasma and its utility in medical dermatology: A systematic review. J Am Acad Dermatol. 2019 Sep;81(3):834-846. doi: 10.1016/j.jaad.2019.04.037. Epub 2019 Apr 19. PMID 31009668
- [Background] Shao S, Pan R, Chen Y. Autologous Platelet-Rich Plasma for Diabetic Foot Ulcer. Trends Endocrinol Metab. 2020 Dec;31(12):885-890. doi: 10.1016/j.tem.2020.10.003. Epub 2020 Nov 13. PMID 33199085